CLINICAL TRIAL: NCT05405257
Title: Oxytocin Treatment for Chronic Pain in Hypermobile Ehlers-Danlos Syndrome
Brief Title: Oxytocin for Hypermobile Ehlers-Danlos Syndrome
Acronym: EDS-OXY
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study team has decided to close the trial (NCT05405257) due problems with patient recruitment and enrollment efforts. To date, only one patient completed both arms.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Brendan Lee, Chairman and Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-45648
Record Dates: First submitted 2022-06-02; First posted 2022-06-06 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Hypermobile Ehlers-Danlos Syndrome; Pain Assessment
Keywords: EDS, Oxytocin, Pain, Hypermobile Ehlers-Danlos Syndrome
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3; Pain | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: This will be a single-blind study. This study will include two treatment periods in a fixed order. One for placebo and one for oxytocin. The participants was blinded to the sequence of treatment assignment which is fixed.
Masking Description: Participant will be blinded to the sequence of treatment (which was fixed). Infusion bags containing either the placebo and drug will not be labeled or known to the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Placebo-Oxytocin sequence (Experimental): In this single blind fixed sequence study participants were treated with Placebo infusion: IV 0.9% NaCl, rate is 200ml over 40 minutes once a day for three consecutive days (one per day) and a after a washout of at least a month Treatment infusion: IV 1IU Oxytocin in 200ml of 0.9% NaCl, rate is 200ml over 40 minutes. Total of three infusions in three consecutive days (one per day)
  Interventions: Drug: Oxytocin; Other: Placebo

INTERVENTIONS:
Drug: Oxytocin — IV 1IU Oxytocin in 200 ml 0.9%NaCl over 40 minutes. Total of three infusions in three consecutive days (one per day).
Other: Placebo — IV, 200 ml 0.9%NaCl over 40 minutes. Total of three infusions in three consecutive days (one per day).

SUMMARY:
The purpose of this pilot study is to evaluate effect of IV oxytocin on chronic pain in patients with Hypermobile Ehlers Danlos syndrome.

DETAILED DESCRIPTION:
This will be a single-site study to evaluate the effect of IV oxytocin on chronic pain in female adult patients with hypermobile EDS.

Oxytocin secretion in the body is dynamic and can be affected by multiple factors including the menstrual period. In order to have minimum variation between tested individuals we conduct this study in females at the same stage of their menstrual cycles. Hypermobile EDS is more prevalent in females and the symptoms are usually more severe in females and more females come to medical attention. We are not aware of any difference in the risk from using oxytocin in females vs males.

All participating individuals are affected with hypermobile-EDS (hEDS) with chronic moderate to severe pain. Study will include two periods of treatment - one with placebo and one with oxytocin and a one month period will be held in between the two treatments. Participants will be blinded to the order of treatment. Each period of treatment will start 7-10 days after the beginning of the menstrual cycle and will include 6 days of daily subjective pain evaluation using pain-evaluation questionnaire ('preinfusion evaluation') followed by three consecutive daily infusions (placebo or oxytocin). Response to treatment will be evaluated by questionnaire during 6 days after each three infusion days (placebo or oxytocin) . Additional questionnaires for evaluation of anxiety and depression will be used as well. Patients will be asked to wear ACTIHEART device (measures heart rate, heart rate variation, and activity levels) 3 days prior to infusion, during the 3 days of infusion, and in the 3 days after the last infusion day. For each infusion period, participants will arrive to the study site for three daily consecutive visits, each will last for 3-4 hours. Response variables will be collected prior, during and after each infusion. Patients will fill out pain evaluation questionnaires pre and post infusion and some questionnaires during the days of infusion. Blood pressure and heart rate measurements will be taken prior, during and after the infusion. Blood samples for measurements of oxytocin levels and blood samples for future analysis will be collected in some of the infusion days (before and after the infusion).

ELIGIBILITY:
Inclusion Criteria:

1) Premenopausal Females, Age >18 years 2) Clinical diagnosis of hypermobile EDS according to the 2017 criteria for hEDS 3) Menstrual periods (range from 8 to 42 days) 4) Pain level greater that pain score of 4 out of 10 on a Numeric Rating Scale in at least two of the following locations: back, neck, shoulders, elbows, wrist, hand joints, hips, knees, ankles, on most days over the 3 months preceding enrollment. 5) On a stable regimen for pain control without any expected increase in dose of pain medications during the study period. 6) All participants should have a negative urine pregnancy test and agree to use an acceptable method of contraception (abstinence or barrier methods).

Exclusion Criteria:

1) Known allergy to OXT or preservatives in the medication 2) Pregnancy 3) Lactation 4) A confirmed clinical diagnosis of autoimmune disorders that lead to joint inflammation and joint pain such as SLE, RA, psoriatic arthritis, ankylosing spondylitis, scleroderma, and enteropathic arthritis 5) History of known cardiac arrhythmias (except for asymptomatic sinus tachycardia and sinus bradycardia) 6) Heart rate persistently greater than 110/min or less than 50 per minute 7) QTC of > 450 ms from EKG (electrocardiogram) test 8) Taking oral or other hormonal contraceptives 9) Individuals with a clinical condition which, in the view of the investigator compromises safety 10) Participating in another interventional study.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 2 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Lee, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a single blinded study with a fixed sequence. The same subject received the placebo and after a washout of at least 30 days later, the treatment with oxytocin.
Groups:
- Placebo First Then Oxytocin: 1. First intervention (15 days) Placebo infusion: IV 0.9% NaCl, rate is 200ml over 40 minutes. Total of three infusions in three consecutive days (one per day)
  2. Washout of 30 days
  3. Second intervention (15 days) Oxytocin treatment: IV 1IU Oxytocin in 200 ml 0.9%NaCl over 40 minutes. Total of three infusions in three consecutive days (one per day).
Period: Overall Study
Arm/Group | Placebo First Then Oxytocin
Started | 2
Completed | 1
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo First Then Oxytocin Sequence: sequence of Placebo-washout-Oxytocin. Placebo infusion: IV 0.9% NaCl, rate is 200ml over 40 minutes. Total of three infusions in three consecutive days (one per day) Washout of 30 days Treatment infusion: IV 1IU Oxytocin in 200ml of 0.9% NaCl, rate is 200ml over 40 minutes. Total of three infusions in three consecutive days (one per day)
Arm/Group | Placebo First Then Oxytocin Sequence
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Participant's Subjective Reported Chronic Pain
Description: Study evaluated maximum pain level by using the Brief Pain Inventory (BPI). Scale range from minimum value of 1 to maximum value of 10. Higher score indicated more pain (worse outcome).
Time Frame: Pain was self reported and documented on days 1, 3, and 5 of the 6 days period prior or after the treatment with oxytocin or with placebo. An average of the three data points pre or post treatment were calculated.
Population: Only one patient completed the sequence
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo-Oxytocine Sequence: Sequence of treatment:
  Placebo infusion: IV 0.9% NaCl, rate is 200ml over 40 minutes. Total of three infusions in three consecutive days (one per day)
  Washout of 1 month
  Oxytocin: IV 1IU Oxytocin in 200 ml 0.9%NaCl over 40 minutes. Total of three infusions in three consecutive days (one per day).
Arm/Group | Placebo-Oxytocine Sequence
Number analyzed (Participants) | 1
score on a scale
  Mean pain levels pre-placebo (mean of values documented on days 1,3,5 of pre treatment period) | 5.3 (1.15)
  Mean pain levels post placebo (mean of values documented on days 1,3,5 of post treatment period) | 2 (1)
  Mean pain levels pre-OXT (mean of values documented on days 1,3,5 of pre treatment period) | 4.3 (0.58)
  Mean pain levels post OXT (mean of values documented on days 1,3,5 of post treatment period) | 6.7 (2.5)

2. Primary Outcome: Change Between Pre and Post Treatment Pain Scores Using the McGill Pain Questionnaire.
Description: Change in the individual's subjective reported pain following treatment with placebo compared to the change in reported pain following treatment with oxytocin as assessed by McGill Pain Questionnaire.
  The McGill questionnaire is a self-report measure that explores both the quality and intensity of pain. Minimum score: is 0 (no pain) and maximum score is 78 (severe pain). Higher score indicates higher level of pain (worse outcome)
Time Frame: Once prior to treatment with placebo OR oxytocin (day 1 of pre-infusion period / 6 days prior to the infusion) and once after treatment with placebo OR oxytocin (day 1 of post-infusion period / 1 day after the infusion)
Population: One patient who completed the entire sequence
Measure: Number; unit: score on a scale
Arm/Group | Placebo-Oxytocin Sequence
Number analyzed (Participants) | 1
score on a scale
  Pain score pre-placebo (value documented on day 1 of pre-infusion period) | 27
  Pain score post placebo (value documented on day 1 of post-infusion period) | 13
  Pain score pre-OXT (value documented on day 1 of pre-infusion period) | 31
  Pain score post OXT (value documented on day 1 of post-infusion period) | 44

3. Primary Outcome: Change in Participant's Subjective Reported Pain
Description: Study evaluated maximum pain level by using the Numerical pain rating scale. Scale range from minimum value of 1 to maximum value of 10. Higher score indicated more pain (worse outcome).
Time Frame: as for outcome 1
Population: Only one patient completed the sequence
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo-Oxytocine Sequence
Number analyzed (Participants) | 1
score on a scale
  Mean pain levels pre-placebo (mean of values documented on days 1,3,5 of pre treatment period) | 3.3 (1.5)
  Mean pain levels post placebo (mean of values documented on days 1,3,5 of post treatment period) | 1.3 (1.5)
  Mean pain levels pre-OXT (mean of values documented on days 1,3,5 of pre treatment period) | 2.7 (1.2)
  Mean pain levels post OXT (mean of values documented on days 1,3,5 of post treatment period) | 1.7 (1.15)

4. Secondary Outcome: Change Between Pre and Post Treatment Anxiety Scores Using the Hospital Anxiety and Depression Scale Questionnaire.
Description: Change in the individual's anxiety following treatment with placebo compared to the change in reported anxiety following treatment with oxytocin as assessed by Hospital anxiety and depression scale The Hospital anxiety and depression scale is a self-report measure to evaluate anxiety and depression. Minimum score is 0 and maximum score is 21. Higher score indicates higher level of anxiety (worse outcome) 0-7: Normal or no anxiety/depression. 8-10: Mild anxiety/depression. 11-14: Moderate anxiety/depression. 15-21: Severe anxiety/depression.
Time Frame: Once prior to treatment with placebo OR oxytocin (day 6 of pre-infusion period / 1 day prior to the infusion) and once after treatment with placebo OR oxytocin (day 6 of post-infusion period / 6 days after the infusion)
Population: One patient who completed the entire sequence
Measure: Number; unit: score on a scale
Arm/Group | Placebo-Oxytocin Sequence
Number analyzed (Participants) | 1
score on a scale
  Anxiety score pre-placebo (value documented on day 6 of pre-infusion period) | 10
  Anxiety score post placebo (value documented on day 6 of post-infusion period) | 13
  Anxiety score pre-OXT (value documented on day 6 of pre-infusion period) | 12
  Anxiety score post OXT (value documented on day 6 of post-infusion period) | 10

5. Secondary Outcome: Change Between Pre and Post Treatment Depression Scores Using the Hospital Anxiety and Depression Scale Questionnaire.
Description: Change in the individual's depression following treatment with placebo compared to the change in reported depression following treatment with oxytocin as assessed by Hospital anxiety and depression scale The Hospital anxiety and depression scale is a self-report measure to evaluate anxiety and depression. Minimum score is 0, maximum score is 21. Higher score indicates higher level of depression (worse outcome) 0-7: Normal or no anxiety/depression. 8-10: Mild anxiety/depression. 11-14: Moderate anxiety/depression. 15-21: Severe anxiety/depression.
Time Frame: as for outcome 4
Population: One patient who completed the entire sequence
Measure: Number; unit: score on a scale
Arm/Group | Placebo-Oxytocin Sequence
Number analyzed (Participants) | 1
score on a scale
  depression score pre-placebo (value documented on day 6 of pre-infusion period) | 0
  depression score post placebo (value documented on day 6 of post-infusion period) | 4
  depression score pre-OXT (value documented on day 6 of pre-infusion period) | 2
  depression score post OXT (value documented on day 6 of post-infusion period) | 2

6. Secondary Outcome: Change Between Pre and Post Treatment Anxiety Scores Using the "State" Part of the State-Trait Anxiety Inventory (STAI) Questionnaire.
Description: Change in the individual's anxiety following treatment with placebo compared to the change in reported anxiety following treatment with oxytocin as assessed by the "state" part of the State-Trait Anxiety Inventory (STAI) questionnaire. The State-Trait Anxiety Inventory (STAI) is a measure of trait and state anxiety. Minimum score is 20 to maximum score is 80. Higher score indicates higher level of anxiety (worse outcome)
Time Frame: as for outcome 4
Population: One patient who completed the entire sequence
Measure: Number; unit: score on a scale
Arm/Group | Placebo-Oxytocin Sequence
Number analyzed (Participants) | 1
score on a scale
  Anxiety score pre-placebo (value documented on day 6 of pre-infusion period) | 59
  Anxiety score post placebo (value documented on day 6 of post-infusion period) | 44
  Anxiety score pre-OXT (value documented on day 6 of pre-infusion period) | 54
  Anxiety score post OXT (value documented on day 6 of post-infusion period) | 50

ADVERSE EVENTS:
Time Frame: 2 months
Description: none was reported
Groups:
- Sequence Placebo-oxytocin: Placebo infusion: IV 0.9% NaCl, rate is 200ml over 40 minutes. Total of three infusions in three consecutive days (one per day)
  One month of washout
  Treatment infusion: IV 1IU Oxytocin in 200ml of 0.9% NaCl, rate is 200ml over 40 minutes. Total of three infusions in three consecutive days (one per day)
  Note: the placebo and the treatment were not defined as separated arms as the same individual received both placebo and after a washout - oxytocin. The decision for this study design was done due to expected low recruitment rate.
Arm/Group | Sequence Placebo-oxytocin
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT05405257/Prot_SAP_000.pdf